CLINICAL TRIAL: NCT05375539
Title: Angelica Herbal Supplement AGN-CognI.Q Acute Dose Safety and Pharmacokinetics (PK) Dose-Response in Prostate Cancer Patients (PK Dose Trial)
Brief Title: AGN-CognI.Q Acute Dose Safety and Pharmacokinetics Dose-Response in Prostate Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Junxuan Lu, Professor, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PSCI-21-173; R01CA260901 (NIH)
Record Dates: First submitted 2022-05-05; First posted 2022-05-16 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: Angelica gigas Nakai; INM 176; pharmacokinetics
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: After the first subject is enrolled, a 14-day waiting period must occur between each subject before the next subject can be enrolled and dosed. If one subject develops a DLT at any dose level, that subject will cease treatment but will continue safety assessments follow-ups. If a second subject develops a DLT at the same dose level, the trial will be stopped and the dose level below will be the MTD. Any subjects who are at higher dose level at the time of 2nd DLT occurrence, will also stop with no further escalation. All subjects will start at the 800 mg dose (visit 2). Each subject will continue to the next week's dose until a DLT has been reached. However, if 2 DLTs occur at the starting 800 mg dose level, trial will be suspended.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AGN-CognI.Q (Experimental): Dose level +1 (800 mg, 4 CognI.Q capsules, Fast at least 2 h before dose and 1 h after) Dose level +2 (1,200 mg, 6 CognI.Q capsules, Fast at least 2 h before dose and 1 h after) Dose level +3 (1,600 mg, 8 CognI.Q capsules, Fast at least 2 h before dose and 1 h after)
  Interventions: Drug: AGN-CognI.Q

INTERVENTIONS:
Drug: AGN-CognI.Q — Herbal dietary supplement products containing/based on AGN alcoholic extracts (including CognI.Q; Decursinol-50TM, GWB78®, Ache Action, Fast-Acting Joint Formula, EstroG-100/Profemin) are marketed in the US for memory enhancement, pain relief and for women's post-menopausal symptom management.
  Other Names: INM®176

SUMMARY:
This study is to obtain acute dose safety and pharmacokinetics/pharmacodynamics (PK/PD) data in a dose-response trial in prostate cancer patients.

DETAILED DESCRIPTION:
The long-term goal of the study is to conduct human clinical trials to test Angelica gigas Nakai (AGN) root alcoholic extract herbal supplement product (AGN-CognI.Q, or CognI.QTM, made with INM®176 proprietary ingredient, Quality of Life Laboratories, Purchase, NY) as a safe and potential efficacious modality for prostate cancer interception akin to secondary prevention to delay hormonal therapy or avoid it entirely after patients have developed recurrent disease following their standard of care (SOC) surgery and radiation curative treatment. The acute dose safety and pharmacokinetics (PK) and pharmacodynamics (PD) information in the target patient population from the current proposed acute PK dose-response trial will inform the optimal design and execution of the longer-term safety and efficacy (phase I/II) trials.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness and ability to give informed consent.
2. Agree to comply with all study procedures and attend all study visits to the best of their ability.
3. Male with age >=40 years.
4. History of prostate cancer diagnosis. Subjects with history of neuroendocrine or small cell prostate cancer will be excluded. Subjects are eligible if meet one or more of the below criteria:

   1. Patients treated forprostate cancer and no detectable disease on imaging and clinical determination are eligible for enrollment, regardless of risk category.
   2. Patients in the low-risk and favorable intermediate-risk groups who are not currently receiving any treatment or have declined any treatment.
5. Not on concurrent androgen deprivation therapy.
6. ECOG performance status 0-2.
7. Life expectancy of greater than 12 months.
8. Subjects must have normal liver and kidney function as defined below:

   * a) total bilirubin within normal institutional limits,
   * b) AST(SGOT)/ALT(SGPT) < 2.5 X institutional upper limit of normal,
   * c) Creatinine within 1.5 ULN of institutional limits OR creatinine clearance > 50 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal.
   * d) Adequate bone marrow function (Hgb ≥ 9.0 g/dL, Platelets ≥ 100 x 109/L, absolute neutrophil count (ANC) of ≥ 1.5 x 109/L), except for subjects with a history of chronic benign neutropenia, where an ANC of ≥ 1.0 x 109/L are eligible.
9. Subjects must agree to use two medically accepted method of contraception and must agree to continue use this method while on the trial and through at least one week after the last dose of study drug. Acceptable methods of contraception include abstinence, barrier method with spermicide, intrauterine device (IUD) known to have a failure rate of less than 1% per year, or steroidal contraceptive (oral, transdermal, implanted, or injected) in conjunction with a barrier method. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post ovulation methods) withdrawal, spermicides only, or lactational amenorrhea are not acceptable methods of contraception.
10. Subjects must stop the CYP3A4 and CYP2C19 strong inhibitors or inducers 2 weeks prior to the start of the study and during the study.
11. Subjects currently taking herbal supplements containing AGN extract, including CognI.Q, Decursinol-50, Ache Action, Fast-Acting Joint Formula, EstroG-100/Profemin must discontinue these or any other supplements containing these products 4 weeks prior to starting study drug.

Exclusion Criteria:

1. Subjects with distant metastatic cancer. Node positive prostate cancer patients are allowed after completion of treatment.
2. Subjects who are receiving chemotherapy, or oral TKI, or immunotherapy (checkpoint inhibitor).
3. Subjects who are receiving any other investigational agents.
4. Uncontrolled intercurrent illness that would limit compliance with study requirements.
5. All vulnerable patient populations.
6. History of New York Heart Association Class III or IV heart failure, history of a myocardial infarction within 6 months, any uncontrolled cardiac arrhythmia, or any other cardiac related problem that would be considered a contraindication for participation in the opinion of the treating physician.
7. Use of androgen deprivation therapy (ADT) or anti-androgen therapy including LHRH agonist, antagonist, GNRH analogs, and antiandrogens.
8. Subjects who are taking Warfarin/Coumadin.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — participant eligibility is based on self-representation of gender identity.
Enrollment: 12 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Electrocardiography (EKG) QTC Interval | 5-6 weeks
  Cardiac safety measured by EKG QT Interval at baseline, at 5 hours (+/-60mins) and 24 h (+/-2hrs) after study drug treatment every study visit (usually weekly) up to 5 weeks
Safety blood lab tests | 5-6 weeks
  CBC diff for hematological safety and CMP for liver and kidney safety at baseline and 24 +/- 2 h after dose and before the next dose level (the latter also serves as baseline for the next dose).

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 4-6 weeks
  PK metrics of decursin (D) and its isomer decursinol angelate (DA) and their metabolite decursinol (DOH) will be measured in blood collected at pre-each dose baseline (0 h labs= baseline), 2h (+/- 30 mins), 3h (+/- 30 mins), 4h (+/- 30 mins), 5h (+/- 30 mins), 6h (+/-30mins), 7h (+/- 30 mins), and 24 h (+/-2hrs) to estimate Peak Plasma Concentration (Cmax).
Plasma Concentration versus time curve (AUC) | 4-6 weeks
  PK metrics of decursin (D) and its isomer decursinol angelate (DA) and their metabolite decursinol (DOH) will be measured in blood collected at pre-each dose baseline (0 h labs= baseline), 2h (+/- 30 mins), 4h (+/- 30 mins), 6h (+/-30mins) and 24 h (+/-2hrs) to estimate Area under the Plasma Concentration versus time curve (AUC).

CONTACTS AND LOCATIONS:
Overall Officials: Monika Joshi, MD, Principal Investigator — Penn State Cancer Institute
Locations (1):
- Penn State Cancer Institute, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All research materials and data, generated by this grant, will be distributed freely or deposited into a repository/stock center making them available to the broader scientific community, either before or immediately after publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year after publication